CLINICAL TRIAL: NCT03813173
Title: Central Cervical Dissection for Clinical Node Negative Papillary Thyroid Carcinoma: a Prospective Study
Brief Title: Central Cervical Dissection for Clinical Node Negative Papillary Thyroid Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Luo Dingcun, vice president of hospital, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangU20190116
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Lymph Node Metastases
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- central cervical dissection (Active Comparator)
  Interventions: Procedure: lymph node dissection
- non central cervical dissection (Experimental)
  Interventions: Procedure: lymph node dissection

INTERVENTIONS:
Procedure: lymph node dissection — The patient was operated under general anesthesia with cervical hyper extension. The affected side or bilateral glandular lobes were resected routinely, which was confirmed as PTC by frozen section. Then one or both central lymph node dissection were separately packed and sent for examination. Scope of lymph node dissection in central carotid region: hyoid bone at the upper border, anonymous artery at the lower border, bilateral common carotid artery at the inner edge, shallow from the superficial layer of deep cervical fascia, deep to the deep layer of deep cervical fascia (anterior fascia). The right recurrent laryngeal nerve (RLN) passes through the central area of the right neck and should be specially protected.

SUMMARY:
This study is divided into three stages. In the first stage, the investigators try to explore the objective clinical imaging standard of cN0PTC on the basis of previous studies, formulate the "clinical imaging standard of cN0PTC", and randomly enroll 2000 patients under the premise of meeting the standard to establish the "predictive model of cN0-pN+PTC".

In the second stage, 2000 patients will be enrolled to test and improve the evaluation efficiency of "cN0-pN+PTC prediction model".

In the third stage, 2 000 patients without lymph node metastasis assessed by "cNo-pN+ PTC prediction model" will be randomly divided into experimental group and control group. The experimental group will be treated with pCND, while the experimental group will be treated without pCND. The central lymph node metastasis probability, the number and size of metastatic lymph nodes in the control group will be observed after operation. The two groups will be followed up for 5, 10, 15 and 20 years to observe the RFS and OS, so as to further evaluate the "cN0-pN+PTC prediction model" scientifically.

ELIGIBILITY:
Inclusion Criteria:

* Phase I and II:

  1. aged 18 to 80 years old;
  2. the primary treatment of patients with unilateral or bilateral PTC;
  3. ultrasound showed that the tumor was localized in the thyroid gland, and the maximum diameter of each lesion was less than 4cm;
  4. ultrasonography of cervical VI lymph nodes: the shortest diameter < 4 mm, no calcification, no cystic change, no local or global echo enhancement;
  5. CT scan of cervical VI lymph nodes: the shortest diameter < 4 mm, no calcification, no cystic change, no enhancement (CT value 40HU or not higher than banded muscle level), no cluster distribution;
  6. patients will voluntarily enter the study after informed consent;

Phase III:

1. aged from 18 to 80 years old;
2. ultrasound showed that the tumor was localized in the thyroid gland, and the maximum diameter of each lesion was less than 4cm;
3. Unilateral or bilateral PTC without lymph node metastasis assessed by "cNo-pN+ PTC prediction model";
4. patients will voluntarily enter the study after informed consent.

Exclusion Criteria:

* (1) patients refused to participate in the study; (2) non first operation patients; (3) Lateral cervical lymph nodes or distant metastasis; (4) Hashimoto's disease; (5) history of neck trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of thyroid cancer | Participants will be followed from the operation to 20 year (maximum)